CLINICAL TRIAL: NCT03985852
Title: Broadening the Reach, Impact, and Delivery of Genetic Services
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: New York University (Other)
Responsible Party: Principal Investigator, Kimberly Kaphingst, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB_00115509
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Risk Reduction Behavior
MeSH Terms: conditions — Neoplasms; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Directed Standard of Care (Active Comparator): Patients receive pre-test genetic counseling and, if relevant, post-test counseling for a negative result from an automated genetics education assistant.
  Interventions: Other: Patient Directed Standard of Care
- Enhanced Standard of Care (No Intervention): Patients receive standard counseling from a genetic counselor.

INTERVENTIONS:
Other: Patient Directed Standard of Care — The pre-test genetic counseling visit will be conducted through access to an automated genetics education assistant accessed through the patient portal. The automated approach will address all the components of the pre-test counseling and contains content designed by the genetic counselors at the University of Utah and NYU. Patients will have the option to contact genetic counselors through the patient portal, by phone, or in person but this will not be required. All results will be reviewed by a genetic counselor. Negative results will be returned by the automated genetics education assistant. Genetic counselors will return results for pathogenic variants and variants of uncertain significance via phone.
  Arms: Patient Directed Standard of Care

SUMMARY:
The purpose of this study is to compare the uptake of genetic testing among patients randomized with two different models of genetic services delivery (a patient-directed model and an enhanced standard of care model) and examine whether the impact on uptake differs by race/ethnicity and rurality. This study will also compare the effect of these delivery models on adherence to cancer prevention and screening recommendations and other patient responses.

DETAILED DESCRIPTION:
Patient Screening: A comprehensive screening algorithm will identify patients with family history data in various sections of the electronic health record (EHR) who meet current genetic testing criteria. Randomization to study arm (Enhanced Standard of Care or Patient-Directed Standard of Care) will be at the level of the primary care clinic.

Enhanced Standard of Care Patients will be offered the opportunity to schedule a pre-test genetic counseling visit. Pre-test counseling includes review of the family history, risk assessment, discussion of the purpose of genetic testing and possible outcomes, implications for insurance coverage, costs, and assessment of psychosocial needs. Patients can opt to proceed with genetic testing during this session. All test results are returned by a genetic counselor by phone or in person based on the patient preference. A copy of the results and a letter with tailored screening recommendations are returned to the primary care provider and patient via the patient portal or mail.

Patient-Directed Standard of Care The pre-test genetic counseling visit will be conducted through access to an automated genetics education assistant accessed through the patient portal of the electronic health record. The automated approach will address all the components of the pre-test counseling and contains content designed by the genetic counselors at the University of Utah and NYU (New York University). Patients will have the option to contact genetic counselors through the patient portal, by phone, or in person but this will not be required. All results will be reviewed by a genetic counselor. Negative results will be returned by the automated genetics education assistant. Genetic counselors will return results for pathogenic variants and variants of uncertain significance via phone. A copy of the results and a letter with tailored screening recommendations will be provided to the patient and primary care provider via the patient portal.

All patients will be offered the option to schedule follow-up appointments in the genetics clinics.

Genetic Testing:

Genetic testing will be performed by Clinical Laboratory Improvement Act (CLIA)- certified, commercial laboratories based on standard clinical practice. Genetic testing will not be required to participate in the research questionnaires.

Research Procedures:

Two follow-up questionnaires will be sent via the patient portal following interaction with genetic counseling:

i. Questionnaire #1: For participant who chose to receive genetic testing, a questionnaire will be sent approximately 4 weeks after their genetic results are returned. Through this questionnaire investigators will assess cognitive (i.e., recall, comprehension, uncertainty, risk perceptions), affective (i.e., test-related distress, positive reactions, decision regret), communication responses (i.e., family, provider), experience with genetic counseling, and sociodemographic characteristics. For those who chose not to test, a questionnaire will be sent approximately 4 weeks after last genetic service contact. In this questionnaire investigators will assess experience with genetic counseling, reason for not testing, decision regret, risk perceptions, and sociodemographic characteristics including numeracy.

ii. Questionnaire #2: A questionnaire will be administered approximately 12 months after last genetic services contact. For those who chose to test, this questionnaire will ask about discussion of their test results with their primary care provider, family members, or others, and self-reported use of cancer screenings. For those who decide not to receive genetic testing, investigators will assess the self-reported use of cancer screenings, whether genetic testing was pursued at another time or through another source, communication with family members, and whether other relatives had received testing.

For any participants who would like to complete questionnaires by telephone, a genetic counseling assistant or research coordinator will administer the questionnaire. Calls will be digitally recorded to allow for analysis of comprehension. Each questionnaire will take about 15 minutes to complete. Participants may also complete the questionnaires by mail if they choose.

In addition to the questionnaires, investigators will examine screenings, care or health procedures related to genetic services recorded in the electronic health record to determine if an impact is made because of participation in genetic services.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English or Spanish

AND

* First degree relative or second degree relative diagnosed with the following regardless of age: Ovarian Cancer, Pancreas Cancer

OR

* First degree relative or second degree relative diagnosed with the following <50 years of age: Breast Cancer, Colorectal Cancer, Endometrial Cancer.

OR

* Three of more relatives on the same side of the family diagnosed with the following clusters of cancer regardless of age:

  * Breast Cancer, Ovarian Cancer, Pancreas Cancer, Prostate Cancer
  * Colorectal Cancer, Endometrial Cancer, Ovarian Cancer, Pancreas Cancer, Urinary tract, Brain, Small intestine
  * Melanoma, Pancreas Cancer

OR

* Ashkenazi Jewish ancestry and family history of Breast Cancer, Ovarian Cancer, Pancreas Cancer, Prostate Cancer.

Exclusion Criteria:

* Patients with a prior cancer diagnosis, other than non-melanoma skin cancer, and/or prior genetic counseling or testing related to hereditary cancer.
* Patients unable to access the patient portal

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3073 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kaphingst, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - NYU School of Medicine, New York, New York
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Bather JR, Goodman MS, Harris A, Del Fiol G, Hess R, Wetter DW, Chavez-Yenter D, Zhong L, Kaiser-Jackson L, Chambers R, Bradshaw R, Kohlmann W, Colonna S, Espinel W, Monahan R, Buys SS, Ginsburg O, Kawamoto K, Kaphingst KA; BRIDGE research team. Social vulnerability and genetic service utilization among unaffected BRIDGE trial patients with inherited cancer susceptibility. BMC Cancer. 2025 Jan 31;25(1):180. doi: 10.1186/s12885-025-13495-4. PMID 39891096
- [Derived] Kaphingst KA, Kohlmann WK, Lorenz Chambers R, Bather JR, Goodman MS, Bradshaw RL, Chavez-Yenter D, Colonna SV, Espinel WF, Everett JN, Flynn M, Gammon A, Harris A, Hess R, Kaiser-Jackson L, Lee S, Monahan R, Schiffman JD, Volkmar M, Wetter DW, Zhong L, Mann DM, Ginsburg O, Sigireddi M, Kawamoto K, Del Fiol G, Buys SS. Uptake of Cancer Genetic Services for Chatbot vs Standard-of-Care Delivery Models: The BRIDGE Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2432143. doi: 10.1001/jamanetworkopen.2024.32143. PMID 39250153
- [Derived] Kaphingst KA, Kohlmann W, Chambers RL, Goodman MS, Bradshaw R, Chan PA, Chavez-Yenter D, Colonna SV, Espinel WF, Everett JN, Gammon A, Goldberg ER, Gonzalez J, Hagerty KJ, Hess R, Kehoe K, Kessler C, Kimball KE, Loomis S, Martinez TR, Monahan R, Schiffman JD, Temares D, Tobik K, Wetter DW, Mann DM, Kawamoto K, Del Fiol G, Buys SS, Ginsburg O; BRIDGE research team. Comparing models of delivery for cancer genetics services among patients receiving primary care who meet criteria for genetic evaluation in two healthcare systems: BRIDGE randomized controlled trial. BMC Health Serv Res. 2021 Jun 2;21(1):542. doi: 10.1186/s12913-021-06489-y. PMID 34078380

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Directed Standard of Care | Enhanced Standard of Care
Started | 1554 | 1519
Completed | 400 | 361
Not Completed | 1154 | 1158

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Directed Standard of Care | Enhanced Standard of Care | Total
Number analyzed (Participants) | 1554 | 1519 | 3073
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (9.9) | 44.1 (9.9) | 43.8 (9.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1149 | 1084 | 2233
  Male | 402 | 428 | 830
  Missing | 3 | 7 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 103 | 101 | 204
  Latinx | 165 | 152 | 317
  White | 1055 | 1039 | 2094
  Other | 85 | 92 | 177
  Missing | 146 | 135 | 281

OUTCOME MEASURES:

1. Primary Outcome: Completion of Genetic Testing From Electronic Health Record
Description: Percentage of patients who decide to receive genetic testing
Time Frame: 1 month following pre-test genetic counseling
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Directed Standard of Care | Enhanced Standard of Care
Number analyzed (Participants) | 1554 | 1519
Participants | 191 | 206

2. Secondary Outcome: Completion of Pre-test Genetic Counseling From Electronic Health Record
Description: Percentage of patients who decide to receive pre-test genetic counseling
Time Frame: 1 month after study invitation
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Directed Standard of Care | Enhanced Standard of Care
Number analyzed (Participants) | 1554 | 1519
Participants | 400 | 361

3. Secondary Outcome: Adherence to Colonoscopy: Questionnaire
Description: Adherence to colonoscopy: questionnaire data
Time Frame: 8 weeks and 13 months from pre-test counseling
Population: Population is participants who completed pre-test genetic services and follow-up questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Directed Standard of Care | Enhanced Standard of Care
Number analyzed (Participants) | 115 | 100
Participants | 17 | 24

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patient Directed Standard of Care | Enhanced Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/1554 | 0/1519
Serious Adverse Events (participants affected / at risk) | 0/1554 | 0/1519
Other Adverse Events (participants affected / at risk) | 0/1554 | 0/1519

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03985852/Prot_SAP_000.pdf